CLINICAL TRIAL: NCT03733379
Title: Clinical, Microbiological and Immunological Evaluation of the Effects of Systemic Probiotics in the Periodontal Treatment
Brief Title: Systemic Probiotics in the Periodontal Treatment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Belén Retamal-Valdes (Other)
Responsible Party: Sponsor-Investigator, Belén Retamal-Valdes, Professor, University of Guarulhos
Organization: University of Guarulhos (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE: 74049717.7.1001.5506
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Periodontitis
Keywords: Periodontitis; Probiotic; Metronidazole; Amoxicillin; Scaling and root planing; Periodontal treatment
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing; Metronidazole; Amoxicillin; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator): Scaling and root planing + Placebos of Metronidazole and Amoxicillin three times a day (TID) for 14 days + placebo lozenges of probiotics two times a day for 90 days.
  Interventions: Procedure: Scaling and root planing; Drug: Metronidazole and Amoxicillin placebos; Dietary Supplement: Probiotic placebo
- Probiotic (Experimental): Scaling and root planing + Placebos of Metronidazole and Amoxicillin three times a day (TID) for 14 days + lozenges of probiotics two times a day for 90 days.
  Interventions: Procedure: Scaling and root planing; Drug: Metronidazole and Amoxicillin placebos; Dietary Supplement: Probiotic
- Antibiotic (Experimental): Scaling and root planing + Metronidazole (400 mg/thrice a day,TID) and Amoxicillin (500 mg/ TID) for 14 days + placebo lozenges of probiotics two times a day for 90 days.
  Interventions: Procedure: Scaling and root planing; Drug: Metronidazole; Drug: Amoxicillin
- Antibiotic + probiotic (Experimental): Scaling and root planing + Metronidazole (400 mg/thrice a day,TID) and Amoxicillin (500 mg/ TID) for 14 days + lozenges of probiotics two times a day for 90 days.
  Interventions: Procedure: Scaling and root planing; Drug: Metronidazole; Drug: Amoxicillin; Dietary Supplement: Probiotic placebo

INTERVENTIONS:
Procedure: Scaling and root planing — SRP will be performed in four to six appointments lasting approximately 1 h each, using manual curettes (Hu-Friedy, Chicago, IL, USA) and ultrasonic device (Cavitron Select SPC, Dentsply professional, York, PA, USA) under local anesthesia. The deep sites will be scaled throughout the first week and treatment of the entire oral cavity will be completed in 14 days.
  Other Names: SRP
Drug: Metronidazole and Amoxicillin placebos — Amoxicillin and metronidazole placebos thrice a day for 14 days (beginning with the first SRP session).
  Arms: Control; Probiotic
Drug: Metronidazole — Metronidazole 400 mg thrice a day for 14 days (beginning with the first SRP session).
  Arms: Antibiotic; Antibiotic + probiotic
Drug: Amoxicillin — Amoxicillin 500 mg thrice a day for 14 days (beginning with the first SRP session).
  Arms: Antibiotic; Antibiotic + probiotic
Dietary Supplement: Probiotic — The probiotic contains 2 different strains of Lactobacillus reuteri: L.reuteri DSM 17938 and L. reuteri ATCC PTA 5289 each at a concentration of 1 x 108 CFU per tablet. It will be used 2 times per day by 90 days.
  Arms: Probiotic
Dietary Supplement: Probiotic placebo — The placebo is identical to the active but without L. reuteri. The two Study Products are identical in taste, texture and shape. It will be used 2 times per day by 90 days.
  Arms: Antibiotic + probiotic; Control

SUMMARY:
The aim of this multicenter randomized clinical trial is to evaluate the clinical, microbiological and immunological effects of probiotics as an adjunct to Scaling and Root Planing alone or in combination with Metronidazole and Amoxicillin in the treatment of periodontitis.

DETAILED DESCRIPTION:
The association of scaling and root planing (SRP) with systemic metronidazole (MTZ) and amoxicillin (AMX) has been advocated as one of the most promising therapeutic protocol for the treatment of advanced periodontitis, since the early 2000's. More recently, probiotics has also been suggested as a promising adjunctive treatment for periodontitis due to their antimicrobial and anti-inflammatory properties. Therefore, the aim of this study is to evaluate the clinical, microbiological and immunological effects of probiotics as an adjunct to SRP alone or in combination with MTZ and AMX in the treatment of periodontitis. In this randomized, double-blind, placebo-controlled trial, subjects with periodontitis will be randomly assigned to receive (i) SRP alone, or combined with: (ii) two probiotics lozenges a day for 90 days (Prob), (iii) 400 of MTZ, plus AMX (500 mg) thrice a day (TID) for 14 days (MTZ+AMX), or (iv) Prob and MTZ+AMX. Subjects will be monitored up to 1 year post-therapy. Nine subgingival plaque samples will be collected at baseline and at 3, 6 and 12 months post-therapy; three samples in each of the following pockets categories: shallow (probing depth [PD]≤3 mm), moderate (PD=4-6 mm) and deep (PD≥7 mm). The microbiological samples will be analyzed by checkerboard DNA-DNA hybridization for 40 bacterial species. Two non-contiguous diseased sites (i.e PD and CAL ≥ 5mm, bleeding and probing [BOP] and no furcation involvement) and two non-contiguous healthy sites (i.e. PD and clinical attachment level [CAL] ≤ 4 mm without BoP and/or marginal bleeding) will be randomly chosen per patient for gingival crevicular fluid (GCF) sampling, from the same sites selected for the microbiological monitoring. Peripheral blood samples will also be collected one week after clinical examination. The GCF and blood samples will be analyzed using a multi-analyte method by means of a 17-multiplex fluorescent bead-based immunoassay for 17 cyto/chemokines. The significance of differences over the course of the study will be sought using repeated measures ANOVA and Tukey multiple comparison tests, and at each time point (among groups) using either ANOVA and Tukey multiple comparison tests or ANCOVA with adjustments for the baseline values. The Chi-square test will be used to compare the differences in the frequency of gender, and to compare the differences in the frequency of subjects achieving the clinical endpoint at 1 year and of self-perceived adverse effects. A stepwise forward logistic regression analysis will be performed in order to investigate the impact of predictor variables on the clinical endpoint for treatment, i.e., "presence of ≤4 sites with PD≥5 mm at 12 months post-therapy (yes/no)". The Number Needed to Treat (NNT) with adjunctive antibiotic in order to obtain treatment success (≤4 sites with PD ≥5 mm) will be calculated. The level of significance will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* ≥30 years of age;
* at least 15 teeth (excluding third molars and teeth with advanced decay indicated for extraction);
* a minimum of 6 teeth with at least one site each with probing depth (PD) and clinical attachment level (CAL) ≥5 mm;
* at least 30% of the sites with probing depth (PD) and clinical attachment level (CAL) ≥4 mm and bleeding on probing (BOP);

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* current smoking and former smoking within the past 5 years;
* systemic diseases that could affect the progression of periodontitis (e.g. diabetes, immunological disorders, osteoporosis);
* scaling and root planing an in the previous 12 months;
* antibiotic therapy in the previous 6 months;
* long-term intake of anti-inflammatory medications;
* need for antibiotic pre-medication for routine dental therapy;
* use of orthodontic appliances;
* extensive dental prosthetic rehabilitation;
* allergy to metronidazole and/or amoxicillin.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects reaching ≤ 4 periodontal sites with probing depth (PD) ≥ 5 mm at 12 months | 12 months

SECONDARY OUTCOMES:
Number of sites with PD ≥ 5 mm. | Baseline, 3, 6 and 12 months
Number of sites with PD ≥ 6 mm. | Baseline, 3, 6 and 12 months
Number of sites with PD ≥ 7 mm. | Baseline, 3, 6 and 12 months
Change in the number of sites with PD ≥ 5 mm. | Baseline, 3, 6 and 12 months
Change in the number of sites with PD ≥ 6 mm | Baseline, 3, 6 and 12 months
Change in the number of sites with PD ≥ 7 mm | Baseline, 3, 6 and 12 months
Mean PD changes in sites with initial PD between 4-6 mm | Baseline - 12 months
Mean PD changes in sites with initial PD ≥ 7 mm. | Baseline - 12 months
Mean CAL changes in sites with initial CAL between 4-6 mm | Baseline - 12 months
Mean CAL changes in sites with initial CAL ≥ 7 mm. | Baseline - 12 months
Full-mouth Probing Depth (mm). | Baseline, 3, 6 and 12 months
Full-mouth Clinical Attachment Level (mm) | Baseline, 3, 6 and 12 months
Percentage of sites with bleeding on probing | Baseline, 3, 6 and 12 months
Percentage of sites with plaque accumulation | Baseline, 3, 6 and 12 months
Percentage of sites with marginal bleeding | Baseline, 3, 6 and 12 months
Occurrence of headache obtained through a questionnaire of adverse effects | 14 days after taking antibiotic
Occurrence of headache obtained through a questionnaire of adverse effects | 90 days after taking probiotic
Occurrence of vomiting obtained through a questionnaire of adverse effects | 14 days after taking antibiotic
Occurrence of vomiting obtained through a questionnaire of adverse effects | 90 days after taking probiotic
Occurrence of diarrhea obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic
Occurrence of diarrhea obtained through a questionnaire of adverse effects. | 90 days after taking probiotic
Occurrence of nausea obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic
Occurrence of nausea obtained through a questionnaire of adverse effects. | 90 days after taking probiotic
Proportions of periodontal pathogenic bacterial species. | Baseline, 3, 6 and 12 months
Counts of periodontal pathogenic bacterial species. | Baseline, 3, 6 and 12 months
Counts of chemokines in the crevicular gingival fluid. | Baseline and 12 months
Counts of chemokines in the peripheral blood samples | Baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Magda Feres, Professor, Principal Investigator — University of Guarulhos
Locations (2):
- Brazil (2):
  - Federal University of Paraná, Curitiba, Paraná
  - University of Guarulhos, Guarulhos, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Feres M, Figueiredo LC, Soares GM, Faveri M. Systemic antibiotics in the treatment of periodontitis. Periodontol 2000. 2015 Feb;67(1):131-86. doi: 10.1111/prd.12075. PMID 25494600
- [Result] Feres M, Soares GM, Mendes JA, Silva MP, Faveri M, Teles R, Socransky SS, Figueiredo LC. Metronidazole alone or with amoxicillin as adjuncts to non-surgical treatment of chronic periodontitis: a 1-year double-blinded, placebo-controlled, randomized clinical trial. J Clin Periodontol. 2012 Dec;39(12):1149-58. doi: 10.1111/jcpe.12004. Epub 2012 Sep 27. PMID 23016867
- [Result] Borges I, Faveri M, Figueiredo LC, Duarte PM, Retamal-Valdes B, Montenegro SCL, Feres M. Different antibiotic protocols in the treatment of severe chronic periodontitis: A 1-year randomized trial. J Clin Periodontol. 2017 Aug;44(8):822-832. doi: 10.1111/jcpe.12721. Epub 2017 Jul 26. PMID 28303587
- [Result] Laleman I, Yilmaz E, Ozcelik O, Haytac C, Pauwels M, Herrero ER, Slomka V, Quirynen M, Alkaya B, Teughels W. The effect of a streptococci containing probiotic in periodontal therapy: a randomized controlled trial. J Clin Periodontol. 2015 Nov;42(11):1032-41. doi: 10.1111/jcpe.12464. Epub 2015 Nov 29. PMID 26427036
- [Derived] Retamal-Valdes B, Teughels W, Oliveira LM, da Silva RN, Fritoli A, Gomes P, Soares GMS, Temporao N, Furquim CP, Duarte PM, Doyle H, Faveri M, Figueiredo LC, Feres M. Clinical, microbiological, and immunological effects of systemic probiotics in periodontal treatment: study protocol for a randomized controlled trial. Trials. 2021 Apr 15;22(1):283. doi: 10.1186/s13063-021-05246-0. PMID 33858486